CLINICAL TRIAL: NCT03996616
Title: Head-up Position, Active Compression-decompression Mechanical Cardiopulmonary Resuscitation and Impedance Threshold Device to Improve Outcomes in Out-of-hospital Cardiac Arrest. A Multicenter Prospective Controlled Quasi-experimental Trial
Brief Title: Head-up Position and High Quality Cardiopulmonary Resuscitation in OHCA
Acronym: GRAVITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GRAVITY
Record Dates: First submitted 2019-06-17; First posted 2019-06-25 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Cardiopulmonary Resuscitation; Head-up position
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Prospective, quasi-experimental, controlled, pre- and post-intervention trial, using a difference-in-differences design and involving two study sites
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): During the pre-intervention period, patients will receive standard CPR in the two study groups. Standard CPR will be performed according to the current guidelines.
  The only changes in current practice for the control will be the monitoring of EtCO2 and cerebral oxymetry as early as possible for the firefighter. ETCO2 will be recorded using a small portable ETCO2 monitor (EMMA, Masimo, USA). EMS first responders will receive a specific training in both group to use, recording, and reporting of ETCO2 value during CPR. This device has CE mark (see related CE mark and user manual). Cerebral oximetry will be recorded using a new small portable device (HR500, Nonin, USA). This device allows using an easy to use adhesive sensor with remote Bluetooth connection to a smartphone sized monitor.
- Assigned Intervention (Active Comparator): During the post-intervention period, patients assigned in the intervention group will receive the evaluated intervention (i.e., HUP and ACD-ITD CPR HUP using the 3 devices in combinations, Elegard, Lucas AD and ITD-16)
  Interventions: Device: Head UP Position; Device: Impedance Threshold Device; Device: New Automated CPR

INTERVENTIONS:
Device: Head UP Position — CPR will be performed manually before the patient is placed on a controlled mechanical elevation device who raises the head and thorax, also known as the head-up position (HUP-Elegard, Minnesota Resuscitation Solutions LLC, USA).
  Rescuers will perform CPR as continuously as possible during the placement of the Elegard, with a <10 second pause in chest compressions during the placement of this device. After performing (LUCAS AD + ITD CPR, see other interventions below) for 2 minutes with the head in the 'flat' position, the Elegard device will be turned on and the head will begin to rise as long as the patient is being treated with the ResQPOD-16 and the LUCAS AD. The head will be elevated to approximately 22 cm from the ground to the back of the occiput.
  Arms: Assigned Intervention
Device: Impedance Threshold Device — An an impedance threshold device ITD-16 (ResQPOD-16, Zoll, USA) will be placed on the patient's airway before the head is elevated.
  Arms: Assigned Intervention
Device: New Automated CPR — Automated CPR will be initiated as soon as feasible using a new automated CPR mechanical compression device that provides full active compression-decompression CPR (LUCAS-AD, Stryker, USA).
  Arms: Assigned Intervention

SUMMARY:
Elevation of the head and thorax, also known as Head-up cardiopulmonary resuscitation (HUP CPR), has been studied extensively in pigs in ventricular fibrillation (VF). HUP combined with active compression decompression and impedance threshold device (ACD+ITD) CPR improves vital organ perfusion and results in a doubling of cerebral perfusion when compared with the same method of CPR in the flat or horizontal plane. HUP CPR enhances the drainage of venous blood from the brain, lowers central venous pressures, reduces intracranial pressures during the decompression phase of CPR, redistributes blood flow through the lungs during CPR, and may reduce brain edema. These mechanisms collectively contribute to improved blood flow and less injury to the brain during CPR. These benefits are due in large part to the effects of gravity on the physiology of HUP CPR. Importantly, HUP CPR is dependent upon a means of generating enough forward flow to adequately pump blood "uphill" to the brain.

In this proposed pilot study, CPR will be performed manually before the patient is placed on a controlled mechanical elevation device (Elegard, Minnesota Resuscitation Solutions LLC, USA). An ITD-16 (ResQPOD-16, Zoll, USA) will be placed on the patient's airway before the head is elevated. Automated CPR will be initiated as soon as feasible using a new automated CPR mechanical compression device that provides full active compression-decompression CPR (LUCAS-AD, Stryker, USA).

The proposed feasibility clinical study will be the first ever to test the fully integrated system of ACD+ITD HUP CPR.

DETAILED DESCRIPTION:
Elevation of the head and thorax, also known as Head-up cardiopulmonary resuscitation (HUP CPR), has been studied extensively in pigs in ventricular fibrillation (VF). HUP combined with active compression decompression and impedance threshold device (ACD+ITD) CPR improves vital organ perfusion and results in a doubling of cerebral perfusion when compared with the same method of CPR in the flat or horizontal plane. HUP CPR enhances the drainage of venous blood from the brain, lowers central venous pressures, reduces intracranial pressures during the decompression phase of CPR, redistributes blood flow through the lungs during CPR, and may reduce brain edema. These mechanisms collectively contribute to improved blood flow and less injury to the brain during CPR. These benefits are due in large part to the effects of gravity on the physiology of HUP CPR. Importantly, HUP CPR is dependent upon a means of generating enough forward flow to adequately pump blood "uphill" to the brain.

Animal studies have shown that HUP CPR must be performed in a specific manner to be effective. For example, conventional standard CPR is insufficient, by itself, for effective HUP CPR. Additional means to enhance circulation are needed, such as concurrent use of the ITD and ACD CPR devices. ACD+ITD CPR alone has been shown to improve hemodynamics and survival with favorable neurologic outcome in several human randomized control trials. Animal studies have shown that HUP CPR is best with the combination of ACD+ITD CPR. Studies have shown that CPR must be initiated before elevating the head. Studies have also shown that HUP CPR is dependent upon the time it takes to elevate the head to the HUP. Elevation of the head and thorax should optimally take place over a 2-minute period of time from a flat position to the maximum head up elevation level in order to optimize cerebral perfusion pressures. Too rapid an elevation of the head and thorax can result in a reduction in cerebral arterial pressure when compared with flat CPR.

In this proposed pilot study, CPR will be performed manually before the patient is placed on a controlled mechanical elevation device (Elegard, Minnesota Resuscitation Solutions LLC, USA). An ITD-16 (ResQPOD-16, Zoll, USA) will be placed on the patient's airway before the head is elevated. Automated CPR will be initiated as soon as feasible using a new automated CPR mechanical compression device that provides full active compression-decompression CPR (LUCAS-AD, Stryker, USA).

The proposed feasibility clinical study will be the first ever to test the fully integrated system of ACD+ITD HUP CPR.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old on enrollment
* Witnessed out-of-hospital cardiac arrest

Exclusion Criteria:

* Obvious pregnancy at inclusion
* Cardiac arrest of traumatic origin (including drowning or hanging)
* Cardiac arrest for which resuscitation seems unjustified (inevitable death, terminally ill irreversible condition, too long duration of cardiac arrest, advance personal directives of no-resuscitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Maximum End-tidal carbon dioxide (ETCO2) | Day 0
  The maximum value of ETCO2 during CPR before ROSC measured after a washout period of 4 positive pressure ventilations (~30 seconds with 30:2 compression: ventilation ratio) will be recorded. ETCO2 value reflects both cardiac output (CO) and pulmonary blood flow, and is an indirect indicator of coronary perfusion pressure during CPR. Levels of ETCO2 > 10-15 mmHg have been correlated with return of spontaneous circulation (ROSC) and survival in both animal and human models of cardiac arrest.

SECONDARY OUTCOMES:
Return of spontaneous circulation (ROSC) | Day 0
  Proportion of patients who's recovered a spontaneous circulation after CPR
Alive at hospital admission | Day 0
  Vital status at hospital admission
Survival to hospital discharge | up to 30 days
  Vital status at hospital discharge
Survival at 30 days | 30 days
  Vital status at 30 days
Neurological functional status | Day 30
  As measured by using the modified Rankin Scale (mRS). A score equal to 0 = no symptoms at all, A score equal to 1 = no significant disability, despite symptoms ; able to carry out all usual duties and activities A score equal to 2 = slight disability ; unable to carry out all previous activities but able to look after own affairs A score equal to 3 = moderate disability ; requiring some help, but able to walk without assistance A score equal to 4 = moderately severe disability ; unable to walk without assistance and unable to attend to own bodily needs without assistance A score equal to 5 = severe disability ; bedridden, incontinent and requiring constant nursing care and attention We considered to a score less or equal to 3 will be considered as favourable neurologic outcome
First recorded rhythm | Day 0
  First recorded rhythm and rhythm recorded by EMS (asystole, ryhtme without pulse, ventricular fibrillation or ventricular tacycardia and spontaneous circulation)
Changes in heart rhythm from ventricular fibrillation (VF) | Day 0
  Proportion of patients who's with changes in heart rhythm from VF to non-VF rhythm and vice versa during the EMS intervention
Signs of life | Day 0
  Presence of agonal respirations and other signs of life (pupillary response, movement during CPR) recorded by ALS
Re-arrest rates | Day 0
  We calculated the proportion of patients who's recovered another cardiac arrest during CPR (supported by ALS and EMS)
Non-invasive arterial O2 | Day 0
  Non-invasive arterial O2 saturation values during CPR recorded by EMS
End-tidal carbon dioxide (ETCO2) after CPR initiation | Day 0
  We compared the difference in ETCO2 values between baseline (i.e., within 2 minutes of CPR initiation) and repeated (i.e., within 4 minutes of CPR initiation) measures during the CPR (recorded by ALS and EMS intervention)
Non-invasive cerebral oximetry (rsO2) | Day 0
  Non-invasive cerebral oximetry (rsO2) values during CPR repeated (i.e., within 4 minutes of CPR initiation) measures recorded by ALS and EMS intervention
Left Ventricular (LV) function | Day 0
  LV function will be measured by echocardiography within 12 hours of ROSC at hospital
Non-invasive measurement of blood pressure | Day 0
  Non-invasive measurement of blood (systolic, diastolic and mean blood pressure) pressure during CPR
Intubation difficulty | Day 0
  Intubation difficulty assessed by the Intubation Difficulty Scale score. Score equal at 0 will be considered to easy intubation, score between 0 and 5 will be considered to slight difficulty, score more than 5 will be considered to moderate to major difficulty and score equal to infinite will be considered to impossible intubation
Neuron specific enolase | Day 0 and 24hours
  Serum Neuron specific enolase was measured at admission and 24h after hospital admission
S100 protein | Day 0 and 24hours
  Serum S100 protein was measured- at admission and 24h after hospital admission
Arterial Blood gases | Day 0
  Arterial blood gases (PaO2 partial pressure of oxygen, PCO2 partial pressure of cardon dioxide, pH, HCO3- bicarbonates and SaO2 oxygen saturation) were measured at hospital admission
Serum lactate concentration | Day 0
  The serum lactate concentration was measured at hospital admission
Serum d-dimer concentration | Day 0 and 24hours
  Serum d-dimer concentration was measured at 4hour and 24 hour after admission
Troponin C serum concentration | Day 0 and 24hours
  Troponin C serum concentration was measured at 4hour and 24 hour after admission
Creatinine concentration | Day 0 and 24hours
  Serum creatinine concentration was measured at 4hour and 24 hour after admission
Transaminases concentration | Day 0 and 24hours
  Serum transaminases concentration (ASAT: aspartate aminotransferases and ALAT: alanine aminotransferases) were measured at 4hour and 24 hour after admission
Imaging | 12 hours
  Head CT will be performed within 12 hours of ROSC. Analysis will include the white to gray matter ratio
End-tidal carbon dioxide between witnessed and unwitnessed cardiac arrest out-of-hospital cardiac arrest | Day 0
  We compared the difference in maximum ETCO2 during CPR between values recorded for witnessed and unwitnessed cardiac arrest
ROSC for witnessed and unwitnessed cardiac arrest | Day 0
  Proportion of patients who's recovered a spontaneous circulation after CPR between witnessed and unwitnessed cardiac arrest
Survival to hospital admission for witnessed and unwitnessed cardiac arrest | Day 0
  Vital status at hospital admission between witnessed and unwitnessed cardiac arrest
Survival to hospital discharge for witnessed and unwitnessed cardiac arrest | Up to 30 days
  Vital status at hospital discharge between witnessed and unwitnessed cardiac arrest
Neurological functional status between witnessed and unwitnessed cardiac arrest | Up to 30 days
  As measured by using the modified Rankin Scale (mRS). A score equal to 0 = no symptoms at all, A score equal to 1 = no significant disability, despite symptoms ; able to carry out all usual duties and activities A score equal to 2 = slight disability ; unable to carry out all previous activities but able to look after own affairs A score equal to 3 = moderate disability ; requiring some help, but able to walk without assistance A score equal to 4 = moderately severe disbility ; unable to walk without assistance and unable to attend to own bodily needs without assistance A score equal to 5 = severe disability ; bedridden, incontinent and requiring constant nursing care and attention We consired to a score less or equal to 3 will be considered as favourable neurologic outcome

CONTACTS AND LOCATIONS:
Overall Officials: Monique Sorentino, Study Director — CHU Grenoble Alpes
Locations (2):
- France (2):
  - SAMU 38, Grenoble, Isère
  - SAMU 54 - CHU Nancy, Nancy, Meurthe-et-Moselle

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be submitted for publication. IPD will be shared with other researcher
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data will be available with no restriction